CLINICAL TRIAL: NCT05063799
Title: Pulmonary Rehabilitation After Pregnancy in COVID-19 Infection: A Case Report
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Halime Sinem Barutçu, Physical Therapist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DrLutfiKirdarCH
Record Dates: First submitted 2021-09-28; First posted 2021-10-01 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: COVID-19 Pneumonia; Pulmonary Rehabilitation; Pregnancy
Keywords: COVID-19, pulmonary rehabilitation, pregnant
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a case included pulmonary rehabilitation program (Experimental)
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — pulmonary rehabilitation programs

SUMMARY:
The 33-month pregnant patient was followed in the gynecology service with the complaint of shortness of breath after receiving the covid positive diagnosis and was transferred to the intensive care unit due to acute respiratory failure. She was intubated in the intensive care unit and the baby was taken by cesarean section. Pulmonary rehabilitation steps to be applied to the patient with long-term intensive care hospitalization will be examined.

DETAILED DESCRIPTION:
After the patient was admitted to the chest diseases service, pulmonary rehabilitation was started. The patient was evaluated before starting pulmonary rehabilitation.

Evaluation parameters; vital signs, shortness of breath, oxygen support, grip force and pinchmeter, fatigue, anxiety and depression, cognitive functions. The pulmonary rehabilitation program will be implemented every day during the hospitalization. The pulmonary rehabilitation program will consist of breathing exercises, strengthening training of upper and lower extremity, exercises in bed, mobilization and reducing oxygen support. The patient will be re-evaluated before discharge.Pulmonary rehabilitation after discharge will continue 2-3 days a week.The patient will be re-evaluated at the 3rd, 6th, 9th and 12th months.

ELIGIBILITY:
Inclusion Criteria:

-pregnant and covid patient

Exclusion Criteria:

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
finger muscle power | 15 second
  Peripheral muscle strength will be measured with a pinchmeter
grip strength | 15 second
  Peripheral muscle strength will be measured with dynamometer

SECONDARY OUTCOMES:
Assessment of cognitive | 10 minutes
  Cognitive will be assessed by Montreal Cognitive Assessment. MoCA Test; a score of 19 to 25 indicates mild cognitive impairment. Scores of between 11 and 21 suggest mild Alzheimer's disease. There is some overlap between this type of dementia and mild cognitive impairment, reflecting the difficulty in using a single test to make this type of diagnosis
Assessment of anxiety and depression | 10 minutes
  Anxiety and depression will be assessed by Hospital Anxiety and Depression Scale.The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Assessment of fatigue | 10 minutes
  Fatigue will be assessed by Functional Assessment of Chronic Illness Therapy. The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued)

CONTACTS AND LOCATIONS:
Locations (1):
- Halime Sinem Barutcu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided